CLINICAL TRIAL: NCT04292106
Title: The Effects of Red Spinach Extract Supplementation on Isometric Strength, Resistance Exercise and Cognitive Performance.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lipscomb University (Other)
Responsible Party: Principal Investigator, Jeremy Townsend, Assistant Professor, Lipscomb University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 092619
Record Dates: First submitted 2020-01-17; First posted 2020-03-02 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2022-01

CONDITIONS: Sports

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo
- Red Spinach Extract (RSE) (Experimental)
  Interventions: Dietary Supplement: Red Spinach Extract (RSE)

INTERVENTIONS:
Dietary Supplement: Red Spinach Extract (RSE) — Oral capsules containing 2g of Red Spinach Extract will be consumed daily for 7 days
  Arms: Red Spinach Extract (RSE)
Dietary Supplement: Placebo — Oral placebo capsules will be taken consisting of maltodrextrin daily for 7 days
  Arms: Placebo

SUMMARY:
Red Spinach is a natural food which is a rich source of nitrates, which are beneficial in hemodynamics, cardiovascular function, and have natural hypotensive and antianginal effects. Red spinach extract has been shown to be beneficial in exercise performance, albeit mostly in aerobic exercise. In a previous study in our lab, we found that dietary nitrate consumption resulted in significantly greater isometric force production in teenage males. However, currently there is little know regarding the effects of dietary nitrate supplementation on isometric strength, resistance exercise and cognitive performance.

DETAILED DESCRIPTION:
This research study is designed to measure the effects of red spinach extract (RSE) on markers of physical and cognitive performance during and following anaerobic exercise.

ELIGIBILITY:
Inclusion Criteria:

* 18-34 years old Participants must have at least 1 year of resistance training experience.
* Free of any physical limitations, medications, and supplements that may affect performance, as determined by a health and activity questionnaire.
* Are free of musculoskeletal injuries
* Are not taking medications that may interfere with study measurements

Exclusion Criteria:

* Participants that cannot take either the RSE or placebo supplement will be excluded, as this will be a double-blind study.
* Furthermore, participants that cannot participate in pre- and post-research testing, and/or those that cannot commit to regular training sessions will be excluded.
* Inability to perform physical exercise (determined by health and activity questionnaire)
* Taking any other nutritional supplement or performance enhancing drug.
* Any chronic illness that causes continuous medical care

Ages: 18 Years to 34 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2019-09-26 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Bench Press Repetitions to Fatiuge | Through study completion, during both treatments (~4 weeks)
  Number of repetitions completed in each set during the acute exercise bout will be recorded and analyzed
Bench Press Power | Through study completion, during both treatments (~4 weeks)
  Power during bench press repetitions will be measured via a linear transducer.
Isometric Mid-thigh pull (IMTP) Peak Force | Through study completion, during both treatments (~4 weeks)
  Peak Force will be measured via dual force plates during a full-body isometric strength test.
Isometric Mid-thigh pull (IMTP) Rate of Force Development | Through study completion, during both treatments (~4 weeks)
  Rate of Force development will be measured via dual force plates during a full-body isometric strength test.

SECONDARY OUTCOMES:
Estimated Muscle Blood Flow via Near-infrared Spectroscopy (NIRS) | Through study completion, during both treatments (~4 weeks)
  Measures of muscle oxygenation of the anterior deltoid will be estimated using a NIRS Device.
Cognitive Performance via Stroop Test | Through study completion, during both treatments (~4 weeks)
  The Stroop Color and Word Test (SCWT) is a neuropsychological test used to assess cognitive performance. This will be administered before and after the fatiguing bench press protocol

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Townsend, PhD, Principal Investigator — Lipscomb University
Locations (1):
- Jeremy Townsend, Nashville, Tennessee, United States